CLINICAL TRIAL: NCT04636242
Title: Photodynamic Therapy for Cutibacterium Acnes (C. Acnes) Decolonization of the Shoulder Dermis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SNAM19G.133
Record Dates: First submitted 2020-10-21; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: C. Acnes; Phototherapy; Postoperative Infection; Arthroscopic Rotator Cuff Repair; Shoulder Surgery
MeSH Terms: interventions — Aminolevulinic Acid; Phototherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Phototherapy Group (Experimental): patient will be instructed to apply 5-aminolevulinic acid HCL topical solution to their shoulder prior to their surgery. 16 minutes before skin incision a blue light will be applied to the area of the shoulder where the 5-ALA was administered
  Interventions: Procedure: Skin Biopsy; Drug: 5 Aminolevulinic Acid + Phototherapy
- Group 2: Control Group (Active Comparator): patient will undergo standard of care surgery
  Interventions: Procedure: Skin Biopsy

INTERVENTIONS:
Procedure: Skin Biopsy — A Biopsy of the skin where the arthroscopic instrument will be placed, will be taken and sent to the microbiology lab for analysis
Drug: 5 Aminolevulinic Acid + Phototherapy — 5 aminolevulinic acid solution will be placed on the skin of the shoulder and the participant will receive Photodynamic therapy on the morning of surgery
  Arms: Group 1: Phototherapy Group

SUMMARY:
This is a prospective, randomized controlled trial to evaluation the ability of 5-aminolevulinic acid HCL topical solution photodynamic therapy to decrease the colonization of Cutibacterium acnes (C. acnes- a bacteria commonly found in the dermis of the skin surrounding the shoulder) in order to decrease postoperative joint infections.

-Aminolevulinic acid (ALA) is a naturally occurring metabolite in the synthesis of pathway of cellular heme production. Adding ALA to bacteria encourages porphyrin production which serve as the immediate precursors to heme production. When these porphyrins are illuminated with blue light at an emission peak of 407-420nm, these metabolites become exothermic and cause internal destruction of the bacterial cells. This therapy does not cause any damage to the mammalian cells, which makes PDT safe for human skin treatment.

ELIGIBILITY:
Inclusion Criteria:

* All male patients (>18) undergoing shoulder arthroscopy)

Exclusion Criteria:

* Female patients
* Patients with active acnes
* Patients who have taken antibiotics within a month of their surgery
* Subjects with psoriatic/eczematous lesions on the shoulder girdle
* Patients on anticoagulant therapy
* Patients who have a known allergy to any of the agents used in the study protocol

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women are being excluded because studies have shown that men have a higher bacterial burden of C. acnes than females. The male predisposition has been linked with the habitat of C. acnes being in the hair follicles and therefore the upper body of males would harbor more of the bacterium than females after shoulder surgery.
Enrollment: 120 (Estimated)
Dates: Start 2019-08-22 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in the number of patients who have microbiological results positive for the bacteria C. acnes after treatment with 5-aminolevulinic acid-photodynamic therapy (ALA-PDT) versus those who were not. | 13 days

SECONDARY OUTCOMES:
Decrease Rate of Postoperative Infection | 3 months
  The change in the incidence of postoperative shoulder infections in participants treated with photodynamic therapy versus participants who were not

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States